CLINICAL TRIAL: NCT01323153
Title: A Phase III, Double-blind, Randomized, Placebo-controlled, Multi-center Study Evaluating the Efficacy and Safety of Dalcetrapib on Lipids, Lipoproteins, Apolipoproteins and Markers of Cardiovascular (CV) Risk in Patients Hospitalized for an Acute Coronary Syndrome (ACS) When Treatment is Initiated Within 1 Week After an ACS (Dal-ACUTE)
Brief Title: A Study of Dalcetrapib in Patients Hospitalized For An Acute Coronary Syndrome (Dal-ACUTE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WC25501
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease | interventions — dalcetrapib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Dalcetrapib (Experimental)
  Interventions: Drug: dalcetrapib
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: dalcetrapib — Oral doses of 600 mg once daily for 20 weeks
  Arms: Dalcetrapib
Drug: placebo — Oral doses of matching placebo to dalcetrapib once daily for 20 weeks
  Arms: Placebo

SUMMARY:
This double-blind, randomized, placebo-controlled, multi-center study will evaluate the safety and efficacy of dalcetrapib in patients hospitalized for an acute coronary syndrome (ACS). Treatment will be initiated within 1 week after the ACS. Patients will be randomized to receive dalcetrapib 600 mg as daily oral doses or matching placebo. The anticipated time on study treatment is 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=45 years of age
* Patients admitted to the hospital for acute coronary syndrome (ACS)
* Patients receiving guideline-based medical and dietary management of dyslipidemia

Exclusion Criteria:

* Symptomatic congestive heart failure (NYHA Class III or IV)
* Clinically significant heart disease requiring coronary artery bypass grafting, cardiac transplantation, surgical valve repair/replacement during the study
* Uncontrolled hypertension
* Uncontrolled diabetes
* Severe anemia
* Concomitant treatment with any other drug raising high-density lipoprotein C (HDL-C; eg niacin, fibrates)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (32):
- United States (5):
  - Pensacola, Florida
  - Saginaw, Michigan
  - Saint Cloud, Minnesota
  - Syracuse, New York
  - Rapid City, South Dakota
- Czechia (10):
  - Chrudim
  - České Budějovice
  - Hradec Králové
  - Jihlava
  - Jindřichův Hradec
  - Prague
  - Semily
  - Teplice
  - Zlín
  - Znojmo
- Netherlands (12):
  - Amsterdam
  - Arnhem
  - Beverwijk
  - Breda
  - Den Helder
  - Eindhoven
  - Gouda
  - Heerlen
  - Nieuwegein
  - Nijmegen
  - Rotterdam
  - Sneek
- United Kingdom (5):
  - Edinburgh
  - Glasgow
  - London
  - Stoke-on-Trent
  - Swansea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dalcetrapib | Placebo
Started | 150 | 150
Completed | 133 | 142
Not Completed | 17 | 8

BASELINE CHARACTERISTICS:
Population: 2 Pt. had no intake of study medication and were excluded from ITT
Groups:
- Total: Total of all reporting groups
Arm/Group | Dalcetrapib | Placebo | Total
Number analyzed (Participants) | 148 | 150 | 298
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (9.77) | 60.7 (10.09) | 60.9 (9.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 68
  Male | 114 | 116 | 230
Region of Enrollment [Number; unit: participants]
  Netherlands | 50 | 52 | 102
  Czechia | 74 | 75 | 149
  United States | 10 | 11 | 21
  United Kingdom | 14 | 12 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in High-density Lipoprotein C (HDL-C) Levels After 4 Weeks of Treatment
Time Frame: 4 weeks
Measure: Least Squares Mean (Standard Error); unit: Percentage raise in HDL-C Levels
Arm/Group | Dalcetrapib | Placebo
Number analyzed (Participants) | 148 | 150
Percentage raise in HDL-C Levels | 43.8 (2.5) | 10.1 (2.5)

2. Secondary Outcome: Similarity in Percent Change From Baseline in High-density Lipoprotein C (HDL-C) Levels After 4 Weeks of Treatment in Studies WC25501 and NC20971
Time Frame: 4 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Percent Change of High-density Lipoprotein C (HDL-C) Treatment Levels After 8, 12 and 20 Weeks of Treatment
Time Frame: 20 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Percent Change From Baseline in Blood Lipid Levels
Time Frame: 20 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Percent Change From Baseline in Lipoprotein Levels
Time Frame: 20 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Percent Change From Baseline in Apolipoprotein Levels
Time Frame: 20 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Safety: Incidence of Adverse Events
Time Frame: 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Dalcetrapib | Placebo
Serious Adverse Events (participants affected / at risk) | 10/148 | 13/150
Other Adverse Events (participants affected / at risk) | 7/148 | 8/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalcetrapib (N=148) | Placebo (N=150)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular Tachicardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Tachicardia (Cardiac disorders) | 1 (1) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Extranodal Marginal Zone B-Cell Lymphoma (Malt Type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectosigmoid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Haemorhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Liver Abscess (Infections and infestations) | 0 (0) | 1 (1)
Mycobacterial Infection (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Dyspnea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Somatoform Disorder Gastrointestinal (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalcetrapib (N=148) | Placebo (N=150)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No